CLINICAL TRIAL: NCT00389714
Title: Phase 2 Clinical Study :Evaluation of the Efficacy of Insoluble Antibacterial Nanoparticles Incorporated Into Commercialy Used Composit Resins as an Esthetic Restoration Material in Children
Brief Title: Clinical Evaluation of Esthetic Restorations Placed in Primary Molars With Composite Resin Enriched With Insoluble Anti Bacterial Nano Particles
Acronym: IABN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 191055nano HMO-CTIL
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2007-12-11 (Estimated); Status verified 2007-12

CONDITIONS: Dental Carious; Dental Filling
Keywords: pedodontics; carious; dental restoration; antibacterial; nanoparticles

INTERVENTIONS:
Device: dental restoration

SUMMARY:
Composite resins are presently among the most popular esthetic restorative materials in dentistry. These materials offer excellent esthetic appearance, allow for conservative cavity preparation and are now becoming widely accepted for clinical use in primary molars 1-23. Despite the improvement of their properties, achieved with better materials and incremental placing techniques, composite resin restorations appear to have still several drawbacks: although similar to amalgam in short terms studies, they have a high long term failure rate, mainly due to discoloration, loss of retention and secondary caries3,11,19, are time-consuming and technique sensitive, lack anti-cariogenic potential and can be amenable to secondary caries at the cervical dentin margins 1, 2.

Continued interest in providing advance in restorative esthetic materials led to the development of new generations of composites. Among the newest material developed is the use of minute amount of nanoparticles which convert composites to possess permanent antibacterial properties.

It is of great interest to observe the clinical behavior of this new material when utilized in clinical practice. Thus the aims of the present in-vivo study are:

1. To evaluate the clinical and radiographic performance of the New Restorative System when placed with adhesive systems in class II restorations of primary molars.
2. To assess, by SEM, the micromorphology of the cervical, buccal and lingual margins of the proximal surfaces of the restored teeth retrieved after exfoliation or extraction.
3. To asses, by means of polarized light microscopy, the integrity of the cervical margins of the same retrieved teeth.

DETAILED DESCRIPTION:
Composite resins are presently among the most popular esthetic restorative materials in dentistry. These materials offer excellent esthetic appearance, allow for conservative cavity preparation and are now becoming widely accepted for clinical use in primary molars 1-23. Despite the improvement of their properties, achieved with better materials and incremental placing techniques, composite resin restorations appear to have still several drawbacks: although similar to amalgam in short terms studies, they have a high long term failure rate, mainly due to discoloration, loss of retention and secondary caries3,11,19, are time-consuming and technique sensitive, lack anti-cariogenic potential and can be amenable to secondary caries at the cervical dentin margins 1, 2.

Continued interest in providing advance in restorative esthetic materials led to the development of new generations of composites. Among the newest material developed is the use of minute amount of nanoparticles which convert composites to possess permanent antibacterial properties.

It is of great interest to observe the clinical behavior of this new material when utilized in clinical practice. Thus the aims of the present in-vivo study are:

1. To evaluate the clinical and radiographic performance of the New Restorative System when placed with adhesive systems in class II restorations of primary molars.
2. To assess, by SEM, the micromorphology of the cervical, buccal and lingual margins of the proximal surfaces of the restored teeth retrieved after exfoliation or extraction.
3. To asses, by means of polarized light microscopy, the integrity of the cervical margins of the same retrieved teeth.

STUDY DESIGN The study will be performed at the Post Graduate Clinic of the Pediatric Dentistry Department of the Hadassah School of Dental Medicine in Jerusalem. The project will have to be approved by the Human Ethical Committee (Helsinki), at the Hadassah Hospital and by the Israeli Ministry of Health.

The study will be double blind, randomized, two-cell, split mouth, design.

The following clinical treating procedures will be tested:

1. Fissure sealants in permanent teeth
2. Class II restorations of primary molars.

A. SUBJECT SELECTION To be eligible to participate in the study the children will have to be between 5 to 10 years old, and present at least two primary molars with a small to moderate proximal carious lesion. These should be in proximal contact with an adjacent tooth and with an antagonist. The children will have to be available for recall appointments every six months until exfoliation of the teeth, and have parental consent to participate in this study.

Following medical history and clinical examination, bilateral bite-wing radiographs will be taken, for diagnosis of caries that need to be restored after assessment of the patient's caries risk 24.

The teeth suitable for the study will be randomly assigned to be restored with one of the two groups:

1. - restoring with commercial composite - hereafter control group
2. - restoring with commercial composite supplemented to which

B. CLINICAL PROCEDURE After local anesthesia, the teeth will be isolated with a rubber dam, and tooth preparation will be made using a #330 carbide bur under water coolant spray, having their cervical margins placed on enamel. Cavity design will be limited to caries removal without an occlusal lock, but grooves will be placed on the occlusal buccal and palatal surfaces. Line and point angles will be rounded (Fig. 1).

Fig 1: demonstrates first and second maxillary primary molars preparations before the insertion of the restorative material.

. Restorative steps

1. Placement of a T-band metal matrix and inserting a wedge firmly, burnishing the matrix band to establish proximal contour and contact area;
2. Acid etching of enamel and dentin for 15 seconds and rinsing;
3. Removal of excess water leaving the surface moist;
4. Appling two layers of Single Bond adhesive to enamel and dentin using a brush saturated with adhesive, and gently drying for 2-5 seconds;
5. Light curing for 10 seconds;
6. Applying the Restorative System incrementally.
7. Curing each increment for 40 seconds;
8. Removal of the band and curing for another 20 seconds from buccal and lingual at the cervical area.

h. Finishing and polishing the restorations using 3M™ ESPE™ Sof-Lex™ Finishing and polishing System.

1. Placement of a T-band metal matrix and inserting a wedge firmly, burnishing the matrix band to establish proximal contour and contact area;
2. Applying Adper Prompt L-Pop to the entire surface of the cavity and rubbing for 15 seconds.
3. Blow dry, light curing for 10 seconds.
4. Applying Filtek™ Supreme Universal Restorative System incrementally.
5. Curing each increment for 40 seconds;
6. Removal of the band and curing for another 20 seconds from buccal and lingual at the cervical area.
7. Finishing and polishing the restorations using 3M™ ESPE™ Sof-Lex™ Finishing and polishing System.

C. EVALUATION

CLINICAL The restorations will be evaluated at baseline- immediately after completion, at six months and yearly thereafter for at least three years, or until tooth exfoliation or patient drop out. The following parameters will be examined: surface appearance, color match, marginal adaptation, marginal discoloration, anatomic form and secondary caries, using the criteria described by Cvar and Ryge (1971)25 -see attached evaluation sheet.

30 restorations of each group will be randomly selected and photographed with a digital camera at baseline and after each follow up examination. The stored photographs will be assessed using the same parameters as for the clinical evaluation.

CONTACT AREA

As part of the clinical evaluation, the quality of the contact area will be assessed with waxed dental floss and classified as follows3:

A. Excellent: resistance was met while passing the dental floss; B. Fair: the contact was present, but the dental floss passed without resistance; C. Poor: No contact existed with the adjacent tooth.

RADIOGRAPHIC EVALUATION Bitewing radiographs will be taken at one-year recall intervals, and will be examined for the presence of radiolucent defects at the cervical margins, and bubbles in the body of the restoration.

POST EXFOLIATION EXAMINATION The patients will be encouraged to bring the teeth to the dental clinic after exfoliation, and they will be promised a financial reward (10.00 ₪-ten Israeli shekels = US$.2.00 approximately). They will be instructed to keep the exfoliated tooth in tap water, and small plastic vials will be provided at the recall examination closest to shedding time. The proximal margins of the retrieved teeth will be evaluated for defects and discoloration using a dental explorer.

SEM EVALUATION OF THE MARGINS

The retrieved teeth will be kept in a humid environment until the time of sectioning. Impressions (Aquasil-Dentsply DeTrey GmbH) will be taken, and epoxy replicas (Epokwick resin, Lake Bluff, IL 60044) of the proximal surfaces will be prepared and gold plated. The micromorphology of the margins will be evaluated by SEM (Jeol JSM 35), and defects at the tooth-restoration interface will be assessed at the cervical proximal margins (buccal and lingual). These defects will be classified according to the fraction of margin length showing gaps wider than 10 microns, as described by Fuks & others 26:

1. No gaps present at the tooth restoration margins;
2. Gaps present at less than 1/3 of the margin;
3. Gaps present at less than 2/3 of the margin;
4. Gaps present along the entire margin.

POLARIZED LIGHT MICROSCOPY The teeth will be embedded in acrylic resin and sectioned following the mesiodistal axis of the tooth, using the Vari/Cut VC-50 sectioning machine (Leco Corp, St. Joseph, MO 49085-2396).

One or two sections of each restoration will be sanded to become thin enough for polarized light examination. The specimens will be examined in water imbibition medium using a polarized light stereomicroscope at X20 magnification. Wall lesions and demineralization areas adjacent to the gingival margins of each restoration will be measured at an enamel distance of 100 microns, a standard distance for most recurrent caries studies27.

D. DATA COLLECTION AND ANALYSIS The restorations, contact areas, radiographs, SEM and polarized microscopy will be evaluated by at least two evaluators. In case of disagreement, the teeth will be reevaluated and the case will be discussed to reach consensus.

The results obtained will be analyzed for statistical differences between the groups.

Table I: Experimental Design: Distribution of the restored teeth.

Group Number of teeth Type of restoration

1. 60 Filtek Supreme + Single Bond Adhesive System
2. 60 Filtek Supreme + Adper Prompt L- Pop

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in the study the children will have to be between 5 to 10 years old, and present at least two primary molars with a small to moderate proximal carious lesion. These should be in proximal contact with an adjacent tooth and with an antagonist. The children will have to be available for recall appointments every six months until exfoliation of the teeth, and have parental consent to participate in this study.

Exclusion Criteria:

* systemic disorders.
* chemotherapy in the last five years

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2007-02

CONTACTS AND LOCATIONS:
Overall Officials: Michael Perez Davidi, DMD, Study Director — Hadassah Medical Organization; Ana Fux, DMD, Study Chair — Hadassah Medical Organization; Mordechay Moskovitch, DMD, Study Director — Hadssah Medical Orgenization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] I -Tonn B and Ryge G: Clinical evaluation of composite resin restorations in primary molars: a 4-year follow-up study. JADA 117:603-606, 1988. 2 -Letzel H: Survival rates and reasons for failure of posterior composite restorations in multicenter clinical trial. JDent 17:S10-S17, 1988. 3- Fuks AB, Araujo FB, Osorio LB, Hadani PE, Pinto AS. Clinical and radiographic assessment of Class II esthetic restorations in primary molars. Pediatr Dent. 2000 Nov-Dec;22(6):479-85. 4 -Yap AU, Chew CL, Ong LF, Teoh SH: Environmental damage and occlusal contact area wear of composite restoratives. J Oral Rehabil. 29:87-97, 2002. 5 -Yap AU, Tan SH, Wee SS, Lee CW, Lim EL, Zeng KY: Chemical degradation of composite restoratives. J Oral Rehabil. 28:1015-21, 2001. 6 -Baratieri LN, Ritter AV: Four-year clinical evaluation of posterior resin-based composite restorations placed using the total-etch technique. J Esthet Restor Dent. 13:50-7, 2001. 7 -Attin T, Opatowski A, Meyer C, Zingg-Meyer B, Buchalla W, Monting JS: Three-year follow up assessment of Class II restorations in primary molars with a polyacid modified composite resin and a hybrid composite. Am J Dent. 14:148-52, 2001. 8 -Kohler B, Rasmusson CG, Odman P. A five-year clinical evaluation of Class II composite resin restorations. J Dent. 28:111-6, 2000. 9 -Pesun IJ, Olson AK, Hodges JS, Anderson GC: In vivo evaluation of the surface of posterior resin composite restorations: a pilot study. J Prosthet Dent. 84:353-9, 2000. 10 -Wang NJ: Is amalgam in child dental care on its way out? Restorative materials used in children and adolescents in 1978 and 1995 in Norway. Community Dent Health. 17:97-101, 2000. 11 -Duncalf WV, Wilson NH: A comparison of the marginal and internal adaptation of amalgam and resin composite restorations in small to moderate-sized Class II preparations of conventional design. Quintessence Int. 31:347-52,2000. 12 -Feigal RJ: Advantages of new restorative materials in dental care for children. J Mich Dent Assoc. 81:32-6, 38, 1999. 13 -Berg JH: The continuum of restorative materials in pediatric dentistry--a review for the clinician. Pediatr Dent. 20:93-100, 1998. 14 -McWhorter AG, Seale NS: For a limited time only! Or treatment of temporary teeth in tots. Tex Dent J. 114:21-6, 1997. 15 -Christensen GJ: Restoration of pediatric posterior teeth. J Am Dent Assoc.127:106-8, 1996. 16 -Croll TP: Restorative dentistry for preschool children. Dent Clin North Am.39:737-70, 1995. 17 -Granath L, Schroder U, Sundin B: Clinical evaluation of preventive and class-I composite resin restorations. Acta Odontol Scand. 1992 Dec; 50(6): 359-64. 18 -Ostlund J, Moller K, Koch G: Amalgam, composite resin and glass ionomer cement in Class II restorations in primary molars--a three year clinical evaluation. Swed Dent J. 16:81-6, 1992. 19 -Barr-Agholme M, Oden A, Dahllof G, Modeer T: A two-year clinical study of light-cured composite and amalgam restorations in primary molars. Dent Mater. 7:230-3, 1991. 20 -Dietschi D, Holz J: A clinical trial of four light-curing posterior composite resins: two-year report. Quintessence Int. 21:965-75, 1990. 21 -Vann WF Jr, Barkmeier WW, Mahler DB: Assessing composite resin wear in primary molars: four-year findings. J Dent Res. 67:876-9,1988. 22 -Leifler E, Varpio M: Proximoclusal composite restorations in primary molars: a two-year follow-up. ASDC J Dent Child. 48:411-6, 1981. 23 -Tonn EM, Ryge G, Chambers DW: A two-year clinical study of a carvable composite resin used as class II restorations in primary molars. ASDC J Dent Child. 47:405-13, 1980 24- Tinanoff N, Douglas JN: Clinical decision -making for caries management in primary teeth. J Dent Edu 65:1133-1142, 2001. 25- Cvar JF and Ryge G: Criteria for the clinical evaluation of dental restorative .materials. USPHS Publication n.790 p244, San Francisco: US Government Printing Office. 26 -Fuks AB, Holan G, Simon H and Levinstein I: Microleakage of class II glass- ionomer-silver restorations in primary molars. Operative Dent 17:62-69, 1992. 27- Fuks AB, Araujo FB, Donly KJ, Cervantes M: Reliability of Different Techniques to Assess Marginal Defects of Class II Restorations in Retrieved Primary Molars: a visual-tactile, SEM, dye penetration and polarized light microscopy study. The Journal of the Israel Dental Association 19:6-16, 2002.
- See also: Michael Perez Davidi — http://www.mypd.co.il